CLINICAL TRIAL: NCT02551965
Title: Nursing Follow up in Geriatric Oncology : Tracking Time of Caregiver Exhaustion Risk
Acronym: TANGO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 6116
Record Dates: First submitted 2015-09-07; First posted 2015-09-16 (Estimated); Last update posted 2020-07-28 (Actual); Status verified 2020-07

CONDITIONS: Exhaustion; Geriatric Disorder
Keywords: Cancer; Patient; Oncology; Caregiver
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Caregiver of cancer patient followed in geriatric oncology (Experimental): caregiver of cancer patient with 70 years old or more, for which a treatment is planned, along with their long term evolution
  Interventions: Other: Phone nursing follow-up

INTERVENTIONS:
Other: Phone nursing follow-up — From the day of geriatric cancer patient's consultation, nurses will identify caregiver and will follow them by phone (caregiver) during 6 months

SUMMARY:
In geriatric oncology, caregivers are submitted to a risk of exhaustion. To investigate the clinical risk factor of exhaustion, the researchers propose to conduct a prospective observational study during 6 months phone follow up of the caregivers. The recruitment will take place during the oncogeriatric assessment consultation.

DETAILED DESCRIPTION:
The primary purpose aim to describe the caregiver of patient with 70 years old or more, suffered from cancer and for which a treatment is planned, along with their long term evolution.

The secondary purposes are to :

* Assess the exhaustion level felt by this caregiver
* Assess the medium delay of caregiver exhaustion apparition
* Relate factors associated to the medium delay of caregiver exhaustion apparition during patient chemotherapy and/or radiotherapy treatment

ELIGIBILITY:
Inclusion Criteria:

* Caregiver of :

  * patient with 70 years old or more, suffered from cancer and receiving specific cancer treatment (chemotherapy or radiotherapy )
  * Patient evaluated in a specific comprehensive oncogeriatric assessment
  * informed patient given a non-opposition form
  * Patient affiliated to a social protection scheme
* Informed consent given by the caregiver

Exclusion Criteria:

* Patient and caregiver under judicial protection
* Caregiver with understanding difficulties with French language
* Psychological, familial, social or geographic conditions that avoid a good clinical trial continuity
* Patient with ≤ 18 years old
* Caregiver and patient with significant cognitive troubles
* Caregiver and patient located in institution during inclusion period

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2016-01; Primary Completion 2023-04 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Standard collection of sociodemographic caregivers features | 6 months
  subjects will be followed for the duration of patient treatment and follow-up in geriatric department, an average of 6 months. The sociodemographic features will be reported during this period, depending on patient disease and caregiver tasks.
Standard collection of economic caregivers features | 6 months
  subjects will be followed for the duration of patient treatment and follow-up in geriatric department, an average of 6 months. The economic features will be reported during this period, depending on patient disease and caregiver tasks.
Standard collection of physical health caregivers features | 6 months
  subjects will be followed for the duration of patient treatment and follow-up in geriatric department, an average of 6 months. The physical health features will be reported during this period, depending on patient disease and caregiver tasks.
Standard collection of psychological health caregivers features | 6 months
  subjects will be followed for the duration of patient treatment and follow-up in geriatric department, an average of 6 months. The psychological health features will be reported during this period, depending on patient disease and caregiver tasks.
Standard collection of caregivers support frequency | 6 months
  subjects will be followed for the duration of patient treatment and follow-up in geriatric department, an average of 6 months. The caregivers support frequency will be reported during this period, depending on patient disease and caregiver tasks.

SECONDARY OUTCOMES:
The exhaustion level felt by caregiver is assessed with Mini-Zarit scale | 6 months
  subjects will be followed for the duration of patient treatment and follow-up in geriatric department, an average of 6 months
Medium delay of caregiver exhaustion apparition is assessed with Mini-Zarit scale | 6 months
  An exhaustion is noticed when caregiver score is ≥ 2 on Mini-Zarit scale. However, the medium delay of caregiver exhaustion apparition is also assessed with an increasing of 2 points from caregiver baseline score on mini-Zarit scale.
  subjects will be followed for the duration of patient treatment and follow-up in geriatric department, an average of 6 months
Factors associated with medium delay of caregiver exhaustion apparition are determined with caregiver and patient features | 6 months
  subjects will be followed for the duration of patient treatment and follow-up in geriatric department, an average of 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Damien HEITZ, MD, Principal Investigator — Strasbourg's University Hospitals - UCROG
Locations (1):
- Unité de Coordination Régionale en Oncogériatrie - Hôpital de Hautepierre, Strasbourg, France